CLINICAL TRIAL: NCT05628064
Title: Prospective, Feasibility Study to Evaluate Performance, Patient Benefits, and Acceptance of a New 1C70 Energy Storage and Return Prosthetic Foot
Brief Title: 1C70 Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Collaborators: Ottobock SE & Co. KGaA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D000002112; CIV-22-08-040306 (Other: European database on medical devices (EUDAMED))
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Amputation
Keywords: amputation; transtibial; prosthetic foot

STUDY DESIGN:
Intervention Model Description: Randomized cross-over controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1C70 to Pro-Flex XC (Experimental): Transtibial amputees randomized to start with 1C70 and cross over to Pro-Flex XC
  Interventions: Device: 1C70; Device: Pro-Flex XC
- Pro-Flex XC to 1C70 (Experimental): Transtibial amputees randomized to start with Pro-Flex XC and cross over to 1C70
  Interventions: Device: 1C70; Device: Pro-Flex XC

INTERVENTIONS:
Device: 1C70 — Investigational energy storage and return prosthetic foot with using novel elastic elements.
Device: Pro-Flex XC — Commercially available carbon-fiber energy storage and return foot used as comparative foot for transtibial amputee subjects.

SUMMARY:
The objective of this study is to characterize the extent of 1C70 meeting the amputees needs in comparison with their everyday and a comparator foot, in regards of daily activities, mobility and balance, as well as quality of life and pain.

ELIGIBILITY:
Inclusion Criteria:

* Person is at least 18 years old.
* Person is a unilateral transtibial amputee with stabilized residual limb.
* Person is a K3 ambulator based on Medicare Functional Classification Level (MFCL) .
* Person has at least 6 months experience in walking with a prosthesis.
* Person is using an energy storage and return (ESR) foot as their primary everyday foot
* Person has a foot size between 22 and 30.
* Person weights with a prosthesis between 50 and 125 kg (foot size 26 - 30), or between 45 and 100 kg (foot size 22 - 25).
* Person wears a prosthesis daily and ≥ 8 hours/day.
* Person is able to walk at least 500 m without having to make a break.
* Person is willing and able to independently provide informed consent.
* Person is willing to comply with study procedures.

Exclusion Criteria:

* Person is pregnant.
* Person is using a hydraulic foot as their primary everyday foot.
* Person is using a sport foot (e.g., Fillauer AllPro, Ottobock Challenger, Össur Flex-Foot Cheetah) as their primary everyday foot.
* Person is using an ESR foot with an integrated vacuum pump (e.g., Ottobock 1C62 Triton Harmony).
* Person has conditions that would prevent participation and pose increased risk (e.g., unstable cardiovascular conditions that preclude physical activity such as walking).
* Person falls ≥ once a week due to the reasons that are not related to prosthesis (e.g., problems with vestibular system).
* Person is not available for study visits during planned study duration.
* Person is participating in another study or intends to participate in another study during this study´s duration.
* Person cannot personally provide their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Extent of meeting amputees prosthetic foot needs: 1C70 vs everyday foot | 2 months after fitting with the last study feet
  The extent of meeting amputees prosthetic foot needs by 1C70 as measured by a single question with a 0 to 10 scale compared to the same score for everyday foot. Higher score correspond with higher extent of meeting amputees prosthetic foot needs.
Extent of meeting amputees prosthetic foot needs: 1C70 vs comparator foot | 2 months after fitting with the last study feet
  The extent of meeting amputees prosthetic foot needs by 1C70 as measured by a single question with a 0 to 10 scale compared to the same score for comparator foot. Higher score correspond with higher extent of meeting amputees prosthetic foot needs.
Change in patient-perceived mobility (PLUS-M) compared to baseline | Baseline measurement vs 2 months after fitting with 1C70
  The change from baseline perception of mobility as measured by the Prosthetic Limb Users Survey of Mobility (PLUS-M) 12-item short form. The PLUS-M questionnaire provides a T-score that ranges from 21.8 to 71.4. Higher PLUS-M scores correspond with greater mobility.
Change in patient-perceived mobility (PLUS-M) compared to the comparator foot | 2 months after fitting with each of the study feet
  The change from baseline perception of mobility as measured by the Prosthetic Limb Users Survey of Mobility (PLUS-M) 12-item short form. The PLUS-M questionnaire provides a T-score that ranges from 21.8 to 71.4. Higher PLUS-M scores correspond with greater mobility.
Highest pain reported: 1C70 vs everyday foot | Baseline measurement vs 2 months after fitting with 1C70
  The level of pain as a highest pain during preceding 7 days reported on a 0 ("No pain at all") to 10 ("the most intense pain imaginable") scale for the following origins: residual limb, sound limb, back, shoulder & neck area, phantom limb pain, while wearing the 1C70 foot compared to the everyday foot.
Highest pain reported: 1C70 vs comparator foot | 2 months after fitting with each of the study feet
  The level of pain as a highest pain during preceding 7 days reported on a 0 ("No pain at all") to 10 ("the most intense pain imaginable") scale for the following origins: residual limb, sound limb, back, shoulder & neck area, phantom limb pain, while wearing the 1C70 foot compared to the coparator foot.

OTHER OUTCOMES:
Change in patient perceived balance confidence (ABC) compared to baseline: 1C70 vs everyday foot | Baseline measurement vs 2 months after fitting with 1C70
  Perception of balance confidence as measured by the Activities-specific Balance Confidence (ABC) Scale. The questionnaire provides a score that ranges from 0 to 100%. Higher scores indicate greater balance confidence.
Change in patient perceived balance confidence (ABC) compared to baseline: 1C70 vs comparator foot | 2 months after fitting with each of the study feet
  Perception of balance confidence as measured by the Activities-specific Balance Confidence (ABC) Scale. The questionnaire provides a score that ranges from 0 to 100%. Higher scores indicate greater balance confidence.
Quality of life as measured by the EQ-5D-5L: 1C70 vs everyday foot | Baseline measurement vs 2 months after fitting with 1C70
  Measure of health status composed of 5 dimensions: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, anxiety and depression. Each dimension is rated on a 5-point scale indicating the level of perceived problems for each dimension (level 1 indicating no problems and level 5 indicating extreme problems). Each health state can potentially be assigned a summary index score based on societal preference weights for the health state. These weights, sometimes referred to as 'utilities', are often used to compute QALYs for use in health economic analyses. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Quality of life as measured by the EQ-5D-5L: 1C70 vs comparator foot | 2 months after fitting with each of the study feet
  Measure of health status composed of 5 dimensions: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, anxiety and depression. Each dimension is rated on a 5-point scale indicating the level of perceived problems for each dimension (level 1 indicating no problems and level 5 indicating extreme problems). Each health state can potentially be assigned a summary index score based on societal preference weights for the health state. These weights, sometimes referred to as 'utilities', are often used to compute QALYs for use in health economic analyses. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Pain interference: 1C70 vs everyday foot | Baseline measurement vs 2 months after fitting with 1C70
  Perception of pain interference on the usual activities as measured by a single question with a 0 ("Does not interfere") to 10 ("Completely interferes") scale.
Pain interference: 1C70 vs comparator foot | 2 months after fitting with each of the study feet
  Perception of pain interference on the usual activities as measured by a single question with a 0 ("Does not interfere") to 10 ("Completely interferes") scale.
Foot preference overall and for use in several specific activities | 2 months after fitting with the last study feet
  Foot preference overall and for use in several specific activities as measured by a questionnaire from the publication of Morgan et al. (Morgan et al. 2018)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Zentrum für Healthcare Technology der Privaten Hochschule Göttingen (ZHT PFH), Göttingen
  - John+Bamberg, Hanover
  - Pohlig Heidelberg, Heidelberg
  - UKM ProTec, Münster
  - Pohlig Nürnberg, Nuremberg
  - Pohlig Traunstein, Traunstein

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Morgan SJ, McDonald CL, Halsne EG, Cheever SM, Salem R, Kramer PA, Hafner BJ. Laboratory- and community-based health outcomes in people with transtibial amputation using crossover and energy-storing prosthetic feet: A randomized crossover trial. PLoS One. 2018 Feb 7;13(2):e0189652. doi: 10.1371/journal.pone.0189652. eCollection 2018. PMID 29414988
- [Derived] Maciejasz P, Budny T, Sauer M, Umari M, Korber J, Ernst J, Altenburg B, Hahn A, Braatz F. User preference and patient benefits of a novel energy storing and return foot: A randomized, cross-over clinical trial. Prosthet Orthot Int. 2025 Dec 1;49(6):645-653. doi: 10.1097/PXR.0000000000000415. Epub 2024 Dec 4. PMID 39630588